CLINICAL TRIAL: NCT01701648
Title: Phase I-II, Randomized, Intraindividually Placebo Controlled Clinical Trial, to Evaluate the Efficacy of Autologous Melanocyte Transplantion on Amniotic Membrane as a Substrate for Patients With Stable Vitiligo.
Brief Title: Melanocyte Transplantation for Patients With Stable Vitiligo.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LEA/VIT; 2009-017757-36 (EudraCT Number)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-09

CONDITIONS: Stable Vitiligo
Keywords: Vitiligo, amniotic membrane, malanocytes, C02 laser.
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Other: Laser CO2

INTERVENTIONS:
Other: Laser CO2 — Transplantation of autologous melanocytes using amniotic membrane as a substrate. Transplantation of suspension of autologous melanocytes.

SUMMARY:
Vitiligo is an acquired skin disease that significantly impacts the quality of life of patients. Medical treatment of vitiligo includes the use of melanocyte transplantation but the results are variable.

This single center, single blind clinical trial comparing another treatment and also no treatment was designed to assess the efficacy of autologous monocyte transplantation in monolayers on a substrate of amniotic membrane for the treatment of stable vitiligo. Patients will receive the two interventions, melanocyte suspension and monolayer on amniotic membrane and will provide an untreated area as a control.

DETAILED DESCRIPTION:
Main Objective:

The main objective is to assess the efficacy of autologous transplantation of monocytes in monolayers grown on a biological substrate of amniotic membrane in the treatment of stable vitiligo. Using a system of digital imaging analysis the percentage of re-pigmentation obtained will be studied after 3, 6 and 9 months of treatment.

Secondary Objectives:

To demonstrate differences in efficacy (as measured by the percentage of re-pigmentation) of each of the 2 techniques used: pure melanocytes in suspension and amniotic membrane with melanocytes in monolayers.

To assess how rapidly epithelialization occurs and the cosmetic result in the short and long term of the areas treated with each of the techniques.

To assess if de-epidermization with CO2 laser may be by itself a stimulus for the reservoir of melanocytes in the adjacent epidermis or hair follicles or if the re-pigmentation obtained with this procedure is merely postinflammatory as a result of trauma to the epidermis.

ELIGIBILITY:
Inclusion criteria

* Patients must voluntarily provide informed consent before any of the tests included in the trial which do not form part of standard treatment can be performed.
* Mentally stable patients, suffering from piebaldism, vitiligo of metameric distribution, focal or generalized vitiligo which has remained stable for at least one year without de-pigmentation or spontaneous re-pigmentation after standard medical treatment.
* A minimum hypopigmented area to treat of 100 cm2 (at least 30 cm2 for each of the therapeutic options).
* For women of child-bearing age, a negative pregnancy test.

Exclusion criteria:

* Women who are pregnant or breast-feeding.
* Positive results in any of the blood tests given
* Concomitant serious illness.
* Patients who have received any agent currently the focus of research in the 30 days prior to their inclusion.
* Patients currently participating in another clinical trial or receiving any other agent currently the focus of research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Autologous Melanocyte Transplantion on Amniotic Membrane as a Substrate for Patients With Stable Vitiligo | six months

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Navarre, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Redondo P, Gimenez de Azcarate A, Nunez-Cordoba JM, Andreu EJ, Garcia-Guzman M, Aguado L, Prosper F. Efficacy of Autologous Melanocyte Transplantation on Amniotic Membrane in Patients With Stable Leukoderma: A Randomized Clinical Trial. JAMA Dermatol. 2015 Aug;151(8):897-9. doi: 10.1001/jamadermatol.2015.0299. No abstract available. PMID 25902042